CLINICAL TRIAL: NCT04984746
Title: Intervention Study With Lettuces Enriched With Iodine and Molybdenum.
Brief Title: Intervention Study on Iodine and Molybdenum Biofortification Vegetables ( Nutri-I-Mo )
Acronym: Nutr-I-Mo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Sara Baldassano, Associate professor, University of Palermo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Nutr-I-Mo-2021
Record Dates: First submitted 2021-07-18; First posted 2021-08-02 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Healthy Diet
Keywords: functional food; Iodine; Molybdenum
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: The study were designed by two cohorts The control group and the interventional group. The intervention lasted for 10 days and 100gr of lettuce per day was consumed.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Intervention: (control group) (Experimental): No Intervention: (control group) The control group was assigned to lettuce without any biofortification but with the same characteristic of bioforticated lettuce(soil, water, harvesting time).
  Interventions: Dietary Supplement: No Intervention: (control group)
- Experimental: intervention group (Experimental): Experimental: intervention group To the intervention group was assigned the biofortificated Molibdenum lettuce and Iodine lettuce.
  Interventions: Dietary Supplement: Experimental: intervention group

INTERVENTIONS:
Dietary Supplement: No Intervention: (control group) — Lettuce without any biofortification was assigned to each participant belonging to the control group which ate 100gr every day for 10 days
  Arms: No Intervention: (control group)
Dietary Supplement: Experimental: intervention group — Molybdenum Iodine group
  Lettuces with Iodine and Molybdenum biofortification was assigned to each participant belonging to the intervention group which ate 100gr of each type of lattuce every day for 10 days
  Arms: Experimental: intervention group

SUMMARY:
The aim of the project is to study the influence of Lettuce crop enriched with Molybdenum and lettuce enriched with Iodine administrated at the same time on healthy population in order to assess influence on hematological parameter and Thyroid hormones. Secondary outcome will be to find out Molybdenum and Iodine presence in urine in order to evaluate vegetables as biocarrier and any additive effect when administrated all together.

DETAILED DESCRIPTION:
Several human pathologies are caused by deficiencies of some mineral elements. These deficiencies can be overcome through careful dietary diversification and mineral supplementation. Increasing the bioavailable mineral concentration in vegetables for human consumption could be a useful tool for prevention of many harmful pathologies. Therefore, in this scenario, it appears very important to identify the right dosages and the most effective methods of administration to bio-fortify vegetables with a strong nutritional-health connotation.

The present project aims to investigate the benefits of fortified food intake in a cohort of healthy individuals. Specifically, participants will be fed with lettuce enriched with Molybdenum and lettuce enriched with Iodine in order to study any additional influence on hematological parameters of both minerals The healthy group will eat 100 gr of Lettuce with iodine and 100gr of lettuce with Molybdenum and collect plasma and urine samples after 10 days. Each subject will be subjected to two venous blood samples taken at the beginning of the observation and at the end. The samples obtained will be transported in certified containers for the safe transport of biological samples, and, subsequently, processed by the experimenters at the laboratories of the Molecular Biology section of the University of Palermo. Serum and plasma will be obtained from each blood sample. All information thus obtained will be recorded in a database in which each person will be identified with a numerical code, in order to comply with current privacy regulations. Body weight, Barefoot standing height, Body mass index, Body composition will be measured in the different groups of study. Samples will be analyzed and compared for glucose, albumin, total cholesterol, HDL-cholesterol, LDL-cholesterol, triglycerides, uric acid, creatinine, AST, ALT, γ-GT, ALP, bilirubin, Ferritin, free Iron, transferrin, total proteins, Magnesium, Calcium, insulin, osteocalcin, hematocrit, hs-CRP, TSH, FT3, FT4. Bone metabolism (Osteocalcin, parathyroid hormone, CTX, Calcitonin), Vitamin D Calcium, Phosphate, Potassium, gastric hormones ( GIP, GLP1, GLP2, ghrelin, glucagon, PYY, CCK) oxidative stress markers (LDL-ox, AGE, urinary 8-iso-prostaglandin F (PGF)2alpha) and inflammatory markers(IL-1, TNF, IL-6, IL-10)

ELIGIBILITY:
Inclusion Criteria:

* Caucasian
* age: 18-65 years
* healthy status
* no drug therapy or integration therapy

Exclusion Criteria:

* Inflammatory chronic disease
* use of medication or suffering from any condition
* pregnancy
* breastfeeding
* current smokers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-04-02 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
Urine Molybdenum and Iodine concentration | 10 days
  Urine Iodine and Molybdenum concentration (mg/l) will be assessed at baseline and after 10 days
Hematology and serum chemistry measurements | 10 days
  (glucose (mg/dL), albumin( mg/dL), total cholesterol (mg/dL), HDL-cholesterol (mg/dL), LDL-cholesterol (mg/dL), triglycerides(mg/dL), uric acid(mg/dL), creatinine(mg/dL), AST (mg/dL), ALT (mg/dL), γ-GT(mg/dL), ALP(mg/dL), Ferritin (mg/dL), free Iron (mg/dL), transferrin (mg/dL), total proteins (mg/dL), Magnesium (mg/dL), Calcium (mg/dL), insulin (mg/dL), Vitamin D (mg/dL), HCRP (mg/dL), Potassium (mg/dL), Phosphate (mg/dL) All these measurements will be assessed at baseline and after 10 days

SECONDARY OUTCOMES:
body mass index (BMI) | 10 days
  Weight (Kg) and Hight (m) will be measured and aggregated to arrive at one reported value. Therefore weight and height will be combined to report BMI (kg/m2)
  All these measurements will be assessed at baseline and after 10 days
body composition | 10 days
  lean mass as percent of body weight and fat mass as percent of body weight will be assessed at baseline and after 10 days
Oxidative stress markers | 10 days
  DL-ox (ng/mL), AGE(ng/mL), urinary 8-iso-prostaglandin F (PGF)2alpha (ng/mL) measured in in plasma will be assessed at baseline and after 10 days
Bone turnover markers | 10 days
  Osteocalcin(ng/L), parathyroid hormone (ng/L), CTX (ng/L), Calcitonin (ng/L) measured in plasma will be assessed at baseline and after 10 days
Gastric hormones | 10 days
  7. GIP (pg/ml), GLP1 (pg/ml), GLP2 (pg/ml), ghrelin (pg/ml), PYY (pg/ml), CCK(pg/ml) measured in plasma will be assessed at baseline and after 10 days
Inflammatory markers | 10 days
  IL-1 (pg/mL), TNF(pg/mL), IL-6(pg/mL), IL-10(pg/mL) measured in plasma will be assessed at baseline and after 10 days

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Biological, Chemical and Pharmaceutical Sciences and Technologies, Palermo University, Palermo, PA, Italy